CLINICAL TRIAL: NCT02703155
Title: The Use of Self-Administered Electronic Oral Glucose Tolerance Test Kit in Screening Cystic Fibrosis Related Diabetes in Children With Cystic Fibrosis
Brief Title: The Use of Home Oral Glucose Tolerance Test Kit in Screening Cystic Fibrosis Related Diabetes
Acronym: HomeOGTT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 14HM13
Record Dates: First submitted 2016-02-09; First posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Cystic Fibrosis Related Diabetes; Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Home Oral Glucose tolerance test kit (Other): Providing children with Cystic Fibrosis between 10 and 17 years of age with Home Oral glucose tolerance test kit to screen Cystic fibrosis related Diabetes.
  Interventions: Device: Home Oral Glucose Tolerance Test kit

INTERVENTIONS:
Device: Home Oral Glucose Tolerance Test kit — Providing Home Oral glucose tolerance test kit to children with Cystic fibrosis for screening Cystic Fibrosis Related Diabetes

SUMMARY:
The aim of this study is to establish if the self-administered electronic Oral Glucose Tolerance Test kit can increase the annual uptake of screening for CFRD in children who are between 10 and 17 years of age with CF.

DETAILED DESCRIPTION:
Cystic fibrosis related diabetes (CFRD) is the most common secondary complication of Cystic fibrosis. It affects nearly 20% of adolescents and 40-50% of adults. Undiagnosed CFRD is associated with significant decline in lung function and nutritional status with an increase in mortality. This emphasises the importance of screening for CFRD in children with CF to minimise the nutritional and pulmonary consequences of diabetes.

The UK CF trust guidelines, the European consensus statement and US Cystic Fibrosis Foundation clinical care guidelines recommend the 2hr (1.75g/kg) oral glucose tolerance test as a screening tool on an annual basis in all CF patients without CFRD.

The American Diabetes Association (A.D.A) recommends that annual screening for CFRD should begin by age 10 years in all CF patients who do not have CFRD. The European Consensus Statement on this is in agreement for screening to start at age 10 years. This standard is often applied within the United Kingdom.

The current gold standard screening tool, the Oral Glucose Tolerance Test, is resource intensive. This requires an individual/child and a parent to attend a clinical facility while fasted and requires trained health care professionals to take venous samples, analyse and interpret the results.

There are also problems encountered in standardising the test. The patient should be fasted and must travel to clinic for the test in the morning. The OGTT, if done at hospital, can therefore affect an individual's time off work, time off school, can cause inconvenience and expensive for an individual, parent and child to travel to clinic. The unpredictability of workload for hospital staff means that test times are often not strictly adhered to or accurately recorded. In patients with cystic fibrosis there is also an additional risk of cross infection when they attend the hospital for OGTT. These factors limit the uptake of OGTTs for screening in children with cystic fibrosis.

To overcome these issues a simple, disposable, self-administered electronic OGTT Kit containing everything required to perform the OGTT at home with simple written and pictorial instructions has been used in this study.

The aim of this study is to establish if the self-administered electronic Oral Glucose Tolerance Test kit can increase the annual uptake of screening for CFRD in children who are between 10 and 17 years of age with CF.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with cystic fibrosis who are between 10 years and 17years old and managed at Great Ormond Street Hospital.

Exclusion Criteria:

* Children who are diagnosed with cystic fibrosis related diabetes.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
proportion of annual screening for Cystic Fibrosis Related Diabetes(CFRD) in children between 10years and 17 years with Cystic Fibrosis(CF) using the Home OGTT device. | 1 year
  Proportion of annual screening for Cystic Fibrosis Related Diabetes(CFRD) in children between 10years and 17 years with Cystic Fibrosis(CF).

SECONDARY OUTCOMES:
User acceptability -Questionnaire | 1 year
  To assess the user acceptability of Home OGTT device.
Variability- timing of sample | 1 year
  To assess if Home OGTT device can reduce the variability of times when the test was done i-e at 0 hrs and 2 hrs later following a glucose drink.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Peters, FRCPCH, MD., Principal Investigator — Great Ormond Street Hospital
Locations (1):
- Great Ormond Street Hospital, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bethel MA, Price HC, Sourij H, White S, Coleman RL, Ring A, Kennedy IE, Tucker L, Holman RR. Evaluation of a self-administered oral glucose tolerance test. Diabetes Care. 2013 Jun;36(6):1483-8. doi: 10.2337/dc12-0643. Epub 2013 Jan 15. PMID 23321216
- [Background] Moran A, Brunzell C, Cohen RC, Katz M, Marshall BC, Onady G, Robinson KA, Sabadosa KA, Stecenko A, Slovis B; CFRD Guidelines Committee. Clinical care guidelines for cystic fibrosis-related diabetes: a position statement of the American Diabetes Association and a clinical practice guideline of the Cystic Fibrosis Foundation, endorsed by the Pediatric Endocrine Society. Diabetes Care. 2010 Dec;33(12):2697-708. doi: 10.2337/dc10-1768. No abstract available. PMID 21115772
- [Background] Wickens-Mitchell KL, Gilchrist FJ, McKenna D, Raffeeq P, Lenney W. The screening and diagnosis of cystic fibrosis-related diabetes in the United Kingdom. J Cyst Fibros. 2014 Sep;13(5):589-92. doi: 10.1016/j.jcf.2014.01.008. Epub 2014 Feb 14. PMID 24529737
- [Background] Management of cystic fibrosis related diabetes mellitus. Report of the UK Cystic Fibrosis Trust Diabetes Working Group; 2004 [June, n.d.].
- [Background] Ode KL, Moran A. New insights into cystic fibrosis-related diabetes in children. Lancet Diabetes Endocrinol. 2013 Sep;1(1):52-8. doi: 10.1016/S2213-8587(13)70015-9. Epub 2013 May 23. PMID 24622267
- [Background] Kern AS, Prestridge AL. Improving screening for cystic fibrosis-related diabetes at a pediatric cystic fibrosis program. Pediatrics. 2013 Aug;132(2):e512-8. doi: 10.1542/peds.2012-4029. Epub 2013 Jul 1. PMID 23821699
- See also: www.diabetes.co.uk — http://www.diabetes.co.uk/oral-glucose-tolerance-test.html